CLINICAL TRIAL: NCT02285751
Title: High "on Treatment" Platelet Reactivity in the Intensive Care Unit
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Bernd Jilma, Ao. Univ.-Prof. Dr. Bernd Jilma, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HTPR-ICU; 2012-002226-76 (EudraCT Number)
Record Dates: First submitted 2012-10-24; First posted 2014-11-07 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Critical Illness
Keywords: high on treatment platelet reactivity; acetylsalicylic acid; clopidogrel; prasugrel; ticagrelor; critically ill; pharmacokinetic; pharmacodynamics
MeSH Terms: conditions — Critical Illness | interventions — Aspirin; Clopidogrel; Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- 200mg acetylsalicylic acid per os (Experimental): patients with high "on treatment" platelet reactivity to acetylsalicylic acid are randomized to 3 different groups, one group receives 200mg acetylsalicylic acid per os
  Interventions: Drug: acetylsalicylic acid
- 100mg acetylsalicylic acid intravenous (Experimental): patients with high "on treatment" platelet reactivity to acetylsalicylic acid are randomized to 3 different groups, one group receives 100mg acetylsalicylic acid intravenously.
  Interventions: Drug: acetylsalicylic acid
- 81 mg chewable acetylsalicylic acid (Experimental): patients with high "on treatment" platelet reactivity to acetylsalicylic acid are randomized to 3 different groups, one group receives 81mg chewable acetylsalicylic acid
  Interventions: Drug: acetylsalicylic acid
- 75mg clopidogrel (Active Comparator): control group for patients with high "on treatment" platelet reactivity to clopidogrel patients continue with standard treatment 75mg clopidogrel/day
  Interventions: Drug: clopidogrel
- 60mg prasugrel (Experimental): Loading dose of prasugrel for patients who remain tested with high "on treatment" platelet reactivity in spite of having received an additional loading dose of 600mg clopidogrel
  Interventions: Drug: prasugrel
- 600mg clopidogrel (Experimental): additional loading dose for 24 patients tested with high "on treatment" platelet reactivity to clopidogrel
  Interventions: Drug: clopidogrel
- 180mg ticagrelor (Experimental): Loading dose of ticagrelor for patients who remain tested with high "on treatment" platelet reactivity in spite of having received an additional loading dose of 600mg clopidogrel Loading dose of ticagrelor for patients who remain tested with high "on treatment" platelet reactivity after being treated with 10mg prasugrel daily
  Interventions: Drug: ticagrelor
- prasugrel 10mg (Active Comparator): patients treated with 10mg prasugrel daily
  Interventions: Drug: prasugrel

INTERVENTIONS:
Drug: acetylsalicylic acid
  Other Names: 100mg Thrombo-ASS; 200mg Thrombo-ASS; 81mg chewable aspirin; 100mg intravenous acetylsalicylic acid
  Arms: 100mg acetylsalicylic acid intravenous; 200mg acetylsalicylic acid per os; 81 mg chewable acetylsalicylic acid
Drug: clopidogrel
  Other Names: 75mg po clopidogrel; 600mg po clopidogrel (loading dose)
  Arms: 600mg clopidogrel; 75mg clopidogrel
Drug: prasugrel
  Other Names: 60mg prasugrel per os loading dose; 10mg prasugrel per os daily
  Arms: 60mg prasugrel; prasugrel 10mg
Drug: ticagrelor
  Other Names: 180mg ticagrelor per os (loading dose)
  Arms: 180mg ticagrelor

SUMMARY:
High "on treatment" platelet reactivity is defined as a poor pharmacodynamic response to the administration of acetylsalicylic acid or clopidogrel. acetylsalicylic acid and clopidogrel are drugs commonly used to reduce platelet activity and prevent cardiovascular events. High "on treatment" platelet reactivity is associated with a higher cardiovascular event rate.

Ticagrelor and prasugrel, like clopidogrel both P2Y12 inhibitors are effective in treating patients with High "on treatment" platelet reactivity to clopidogrel.

Critically ill patients are a unique population with altered pharmacokinetic and pharmacodynamic properties. Gastrointestinal dysmotility with associated altered resorption and impaired microvascular function occur frequently in critically ill patients and may lead to altered resorption of orally administered drugs.

The investigators will test a minimum of 100 patients treated with 100mg acetylsalicylic acid per os and 100 patients treated with 75mg clopidogrel per os to calculate the prevalence of high "on treatment" platelet reactivity.

30 patients with high "on treatment" platelet reactivity to acetylsalicylic acid will be randomized to three new treatment groups. In the first group patients will receive 200mg acetylsalicylic acid per os, in the second group 100mg acetylsalicylic acid intravenously and in the third group 81mg chewable acetylsalicylic acid. Each group will contain 10 patients. Pharmacokinetics and pharmacodynamics will be reassessed to evaluate the new treatment.

36 patients with high "on treatment" platelet reactivity to clopidogrel will be randomized to receive either an additional loading dose of 600mg clopidogrel (n=24) or to continue normal treatment as a control group (n=12). Pharmacokinetics and pharmacodynamics will be reassessed and those patients, who are tested again to have high "on treatment" platelet reactivity in spite of the additional loading dose, will now be randomized to receive either ticagrelor or prasugrel. The investigators expect about six patients per group. The twelve patients in the control group will continue normal treatment (75mg/day) until the end of the study. Pharmacokinetics and pharmacodynamics of ticagrelor and prasugrel will be assessed. Any patient, who is tested again with high "on treatment" platelet reactivity in spite of receiving prasugrel or ticagrelor, will be finally switched to the opposite drug and a final high "on treatment" platelet reactivity testing will be conducted.

16 patients who are treated with 10mg prasugrel per os will be tested for HTPR and if positively tested will be switched to 2x90mg ticagrelor per os per day. Platelet reactivity will be reassessed to test whether switching the medication benefits the patients.

ELIGIBILITY:
Inclusion Criteria:

* >18years of age
* admittance to an intensive care unit

Exclusion Criteria:

* recent surgery
* active bleeding
* known coagulation disorders
* discretion of the physician
* terminal illness (anticipated life expectancy < 3months; e.g. due to cancer)
* pregnancy
* <20000 platelets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-11; Primary Completion 2020-07 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
pharmacodynamics (Arachidonic acid induced aggregation test with multiplate electrode aggregometry) | on average 3 days
  Arachidonic acid induced aggregation test with multiplate electrode aggregometry of patients with high "on treatment" platelet reactivity to acetylsalicylic acid after receiving new treatments as explained.
  adenosine diphosphate induced aggregation tested with multiplate electrode aggregometry of patients with high "on treatment" platelet reactivity to clopidogrel after an additional loading dose clopidogrel, or after receiving prasugrel or ticagrelor

SECONDARY OUTCOMES:
Prevalence of high "on-treatment" platelet reactivity in the intensive care unit | maximum 2 weeks after admission
  percentage of patients tested with high "on treatment" platelet reactivity according to defined values
Evaluation of pharmacokinetics (Serum levels of Salicylate/acetylsalicylic acid, clopidogrel-active metabolite, prasugrel-active metabolite, ticagrelor active-metabolite) | on average 3 days
  Serum levels of Salicylate/acetylsalicylic acid, clopidogrel-active metabolite, prasugrel-active metabolite, ticagrelor active-metabolite
intensive care unit mortality | maximum 90 days
  discharge of ICU
comparison of hemodynamically stable vs unstable ((defined by serum lactate>2.1mmol/l, need for circulatory support) | maximum 3 days
  hemodynamically stable vs unstable (defined by serum lactate>2.1mmol/l, need for circulatory support)
major bleeding (defined by TIMI-TRITON-38 criteria) | average of 2 weeks within inclusion
  assessment of major bleeding incidences defined by TIMI-TRITON-38 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Jilma, Ao. Univ.-Prof. Dr. med, Principal Investigator — Medical University of Vienna, Department of Clinical Pharmacology
Locations (1):
- General Hospital, Vienna, Austria